CLINICAL TRIAL: NCT05099393
Title: Effect of Non-nutritive Sweeteners on Vascular Function in Humans
Acronym: SOSweet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 38RC19.355
Record Dates: First submitted 2021-09-29; First posted 2021-10-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Non Nutritive Sweeteners Consumption
MeSH Terms: interventions — Non-Nutritive Sweeteners

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, controlled, randomized, double-blind, three-period crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subject with obesity (Experimental): composed of subject with obesity (Body mass index > 30)
  Interventions: Dietary Supplement: Non Nutritive Sweeteners
- lean subject (Experimental): composed of healthy volunteers (Body mass index < 30)
  Interventions: Dietary Supplement: Non Nutritive Sweeteners

INTERVENTIONS:
Dietary Supplement: Non Nutritive Sweeteners — The 2 arms will participate in 3 periods and each of these periods will correspond to the intake of either sucralose, AceK or a placebo.
  The order will be defined randomly. There will be 3 periods and each period will last 4 weeks. 7 to 14 days of break will be respected between each period.

SUMMARY:
In recent decades, low-to-null caloric, non-nutritive sweeteners (NNS) have been increasingly used, replacing and offering an alternative to food and beverages sweetened by high-energy, added sugars. Indeed, by providing consumers with products that have a sweet taste with low energy content, NNS appear to be the magic bullet to enhance weight loss and reduce cardio-metabolic diseases. However, a recent meta-analysis of randomized trials does not show any benefit of NNS consumption on body weight loss. Moreover, epidemiological, descriptive and experimental studies have recently reported that NNS consumption is paradoxically associated with weight gain, glucose intolerance and increased risk of type 2 diabetes and/or cardiovascular events. Among the approved NNS, sucralose and AceK, both high intensity (respectively ~500-600 and 200 times sweeter than sugar) are the most widely used in foods and drinks, accounting more than 62 % of the global artificial sweetener market. Recent experimental data show an effect of sucralose and AceK (and other NNS) consumption on vascular reactivity in response to a physiological stress (hyperglycemic load) in rats. Since sweet taste receptors (T1R) have been recently found in the endothelium, investigators hypothesize that NNS, and especially sucralose and AceK, a potent T1R agonist, impairs micro- and macrovascular reactivity in humans, which, to the best of our knowledge, has never been explored.

DETAILED DESCRIPTION:
In recent decades, low-to-null caloric, non-nutritive sweeteners (NNS) have been increasingly used, replacing and offering an alternative to food and beverages sweetened by high-energy, added sugars. Indeed, by providing consumers with products that have a sweet taste with low energy content, NNS appear to be the magic bullet to enhance weight loss and reduce cardio-metabolic diseases. However, a recent meta-analysis of randomized trials does not show any benefit of NNS consumption on body weight loss. Moreover, epidemiological, descriptive and experimental studies have recently reported that NNS consumption is paradoxically associated with weight gain, glucose intolerance and increased risk of type 2 diabetes and/or cardiovascular events. Among the approved NNS, sucralose and AceK, both high intensity (respectively ~500-600 and 200 times sweeter than sugar) are the most widely used in foods and drinks, accounting more than 62 % of the global artificial sweetener market. Recent experimental data show an effect of sucralose and AceK (and other NNS) consumption on vascular reactivity in response to a physiological stress (hyperglycemic load) in rats. Since sweet taste receptors T1R have been recently found in the endothelium, investigators hypothesize that NNS, and especially sucralose and AceK, a potent T1R agonist, impairs micro- and macrovascular reactivity in humans, which, to the best of our knowledge, has never been explored.

This is a prospective, single-center, controlled, randomized, double-blind, three-period crossover study

The principal objective is to evaluate the effect of a NNS daily consumption (sucralose or AceK) during 4 weeks on macrovascular endothelial function, in lean and obese subjects compared to placebo.

The principal outcome / endpoint will be based on flow-mediated dilation (FMD) of the brachial artery, expressed as a percent change from baseline diameter, and corrected for shear rate, according to current recommendations, after 4 week of NNS (sucralose or AceK) daily consumption compared to placebo

CONDUCT OF THE RESEARCH : Patients will be screened and, if eligible, proposed a 3-period crossover trial (sucralose, AceK, placebo). The order will be randomized. These 3 periods will be separated with wash out periods between one and two weeks. The 3 periods of 4 weeks will be with one visit at the beginning and at the end of each period, i.e. a total of 6 visits. During each beginning and end of period visit, microvascular and macrovascular reactivity tests will be conducted. At the first visit only, microdialysis will be performed.

Number of subjects : 40 Length of the inclusion period: 24 months Length of treatment: 3 one-month periods, and maximum 4 weeks of wash-outs Length of participation for each subject: 4 months Total length of the study (with statistical analysis): 36 months

STATISTICAL ANALYSIS ; The analysis of the primary outcome will be carried on using an analysis of covariance (ANCOVA), adjusted on baseline FMD, with a risk alpha of 0.05 and a power of 80%, two-sided. Investogators estimated within-subject correlation to be close to 0.7, as shown in previous results by our group.5 In order to maximise power, for secondary objectives, the effects of sucralose, AceK, sex, and obesity, will be assessed using mixed-effects models, with the subject as a random factor.

EXPECTED IMPACT : This is a hot topic since recent studies in animals and humans do not support the claims previously submitted to regulatory agencies that NNS, including sucralose and AceK, are stable compounds that are not metabolized in vivo; and have no effect on metabolism. Questioning the physiological inactivity of these extensively used molecules is mandatory since there is a rise in the consumption of NNS-containing products. Moreover, very recent studies are observing an increase in the consumption of diet products, especially in vulnerable groups (obese, diabetic patients, children or pregnant women). New data on the effect of chronic NNS consumption will help revisit the regulatory status of NNS and bring extensive knowledge on the role of T1R receptors on vascular function, which has been hardly ever studied so far. Finally and importantly, vascular function is largely recognized as a strong precursor of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged≥ 18 years
* Signed informed consent
* Body mass index:

  * 25 kg/m² ≥ BMI ≥ 18,5 kg/m² (lean subjects)
  * >30 kg/m2, with waist-to-hip ratio >0.9 (subjects with obesity)
* Person who is affiliated to a social security scheme or who is a beneficiary of such a scheme

Exclusion Criteria:

* Any chronic disease with vascular impact (including type 2 diabetes)
* Active tobacco use (any quantity)
* Participant involved in another interventional clinical study
* History of hypersensitivity reaction to products used
* The persons mentioned in articles L1121-5 to L1121-9 of the public health code may not be included in this research (Pregnancy or Lactation ; Females with childbearing potential, defined as a premenopausal female and not using an effective form of birth control. (Effective birth control methods include: oral, implant or patch hormone contraception; intrauterine device; abstinence and outercourse; tubal ligation; vasectomy.) ; Person deprived of liberty by judicial order ; Person under guardianship or curatorship ; Minors ; Adults who are incapable or unable to give their consent ; Cross-over situations)
* Subject who would receive more than 4500 euros in compensation due to his or her participation in other research involving the human person in the 12 months preceding this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Macrovascular endothelial function | through study completion, an average of 4 months
  Flow-mediated dilation (FMD) of the brachial artery, expressed as a percent change from baseline diameter, and corrected for shear rate, according to current recommendations,6 after 4 week of NNS (sucralose or AceK) daily consumption compared to placebo.

SECONDARY OUTCOMES:
Macrovascular non-endothelial function | through study completion, an average of 4 months
  Nitrate-mediated dilation (NMD), expressed as a percent change from baseline diameter, and corrected on the shear rate, in accordance with guidelines, after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Macrovascular endothelial function | through study completion, an average of 4 months
  Flow-mediated dilation (FMD) of the brachial artery, expressed as a percent change from baseline diameter, and corrected on the shear rate, in accordance with guidelines, in response to a glycemic stress, after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Macrovascular non endothelial function | through study completion, an average of 4 months
  Nitrate-mediated dilation (NMD) of the brachial artery, expressed as a percent change from baseline diameter, and corrected on the shear rate, in accordance with guidelines, in response to a glycemic stress, after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Microvascular endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to iontophoresis of acetylcholine (ACh), measured with laser speckle contrast imaging (LSCI), after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Microvascular non endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to iontophoresis of sodium nitroprussiate (SNP), measured with laser speckle contrast imaging (LSCI), after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Microvascular endothelial and non endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to local thermal heating, measured with laser speckle contrast imaging (LSCI), after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Microvascular endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to iontophoresis of acetylcholine (ACh), measured with laser speckle contrast imaging (LSCI), in response to a glycemic stress, after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Microvascular non endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to iontophoresis of sodium nitroprussiate (SNP), measured with laser speckle contrast imaging (LSCI), in response to a glycemic stress, after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Microvascular endothelial and non endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to local thermal hyperheamia, measured with laser speckle contrast imaging (LSCI), in response to a glycemic stress, after 4 weeks of NNS (sucralose or AceK) daily consumption compared to placebo.
Macrovascular endothelial function | through study completion, an average of 4 months
  Flow-mediated dilation (FMD) of the brachial artery, expressed as a percent change from baseline diameter, and corrected on the shear rate, in accordance with guidelines 2 hours after an acute intake of NNS (sucralose or AceK) compared to placebo
Macrovascular non endothelial function | through study completion, an average of 4 months
  Nitrate-mediated dilation (NMD) of the brachial artery, expressed as a percent change from baseline diameter, and corrected on the shear rate, in accordance with guidelines 2 hours after an acute intake of NNS (sucralose or AceK) compared to placebo
Microvascular non endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to iontophoresis of SNP, measured with laser speckle contrast imaging (LSCI), one hour and a half after an acute intake of NNS (sucralose or AceK) compared to placebo.
Microvascular endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to iontophoresis of Ach, measured with laser speckle contrast imaging (LSCI), one hour and a half after an acute intake of NNS (sucralose or AceK) compared to placebo.
Microvascular endothelial and non endothelial function | through study completion, an average of 4 months
  Microvascular reactivity to local thermal hyperhemia measured with laser speckle contrast imaging (LSCI) one hour and a half after an acute intake of NNS (sucralose or AceK) compared to placebo.
Metabolic function | through study completion, an average of 4 months
  Plasma levels of ghrelin, after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Metabolic function | through study completion, an average of 4 months
  Plasma levels of gastric inhibitory peptide (GIP), after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Metabolic function | through study completion, an average of 4 months
  Plasma levels of glucagon like peptide (GLP-1), after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Metabolic function | through study completion, an average of 4 months
  Plasma levels of peptide tyrosine tyrosine (PYY), after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Metabolic function | through study completion, an average of 4 months
  Plasma levels of cholecystokinin (CCK), after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Metabolic function | through study completion, an average of 4 months
  Plasma levels of leptin after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Metabolic function | through study completion, an average of 4 months
  Glycaemia, after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Metabolomics profiles | through study completion, an average of 4 months
  Plasma metabolomics profile after 4 weeks daily consumption of NNS (sucralose or AceK) compared to placebo.
Microvascular and macrovascular endothelial and non endothelial function | through study completion, an average of 4 months
  Results of FMD, NMD, local thermal hyperaemie (LTH) and iontophoresis of Ach and SNP compared between lean and obese subjects, in response to an acute or daily consumption of NNS (sucralose or AceK) or placebo.
Microvascular and macrovascular endothelial and non endothelial function | through study completion, an average of 4 months
  Results of FMD, NMD, LTH, and iontophoresis of Ach and SNP, compared between male and female subjects, in response to an acute or daily consumption of NNS (sucralose or AceK) or placebo.
Microvascular and macrovascular endothelial and non endothelial function | through study completion, an average of 4 months
  Results of FMD, NMD, LTH and iontophoresis of Ach and SNP, according to the basal consumption of sweetener, in response to an acute or daily consumption of NNS (sucralose or AceK) or placebo.
Microdialysis reactivity | First visit, one day
  Microvascular reactivity by microdialysis of sucralose measured with laser speckle contrast imaging (LSCI)
Microdialysis reactivity | First visit, one day
  Microvascular reactivity by microdialysis of AceK measured with laser speckle contrast imaging (LSCI)
Microdialysis reactivity | First visit, one day
  Microvascular reactivity by microdialysis of lactisole measured with laser speckle contrast imaging (LSCI)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu ROUSTIT, Pr, Principal Investigator — Centre hospitalier universitaire grenoble alpes
Locations (1):
- Grenoble University hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
Data can be requested by contacting Prof. Roustit mroustit@chu-grenoble.fr
Supporting Information: Study Protocol